CLINICAL TRIAL: NCT02200718
Title: A Phase I Study of NeuroVax™, a Novel Therapeutic TCR Peptide Vaccine for Pediatric Multiple Sclerosis
Brief Title: A Study of NeuroVax™, a Novel Therapeutic TCR Peptide Vaccine for Pediatric Multiple Sclerosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Immune Response BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR902-007
Record Dates: First submitted 2014-07-17; First posted 2014-07-25 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis Pediatric MS NeuroVax Vaccine Therapeutic
MeSH Terms: conditions — Multiple Sclerosis | interventions — NeuroVax vaccine; HIV-1 immunogen, incomplete Freund's adjuvant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NeuroVax (Experimental): NeuroVax consists of a Trivalent TCR Peptide Formulation in IFA V Beta Peptides BV5S2, BV6S5 and BV13S1 emulsified in incomplete Freund's adjuvant
  Interventions: Biological: NeuroVax
- IFA Incomplete Freund's Adjuvant (Placebo Comparator): IFA Incomplete Freund's Adjuvant is a vaccine adjuvant composed of a light mineral oil a surfactant system designed to make a water-in-oil emulsion
  Interventions: Biological: IFA Incomplete Freund's Adjuvant

INTERVENTIONS:
Biological: NeuroVax — NeuroVax consists of a Trivalent TCR Peptide Formulation in IFA BV5S2, BV6S5 BV13S1
  Other Names: IR902 TCR Peptide Formulation in IFA BV5S2, BV6S5 BV13S1
  Arms: NeuroVax
Biological: IFA Incomplete Freund's Adjuvant — IFA Incomplete Freund's Adjuvant is a vaccine adjuvant composed of a light mineral oil and a surfactant system designed to make a water-in-oil emulsion
  Arms: IFA Incomplete Freund's Adjuvant

SUMMARY:
A Phase I Study of NeuroVax™, a Novel Therapeutic TCR Peptide Vaccine for Pediatric Multiple Sclerosis to demonstrate safety & efficacy

DETAILED DESCRIPTION:
A Multi-Center Phase I Study of NeuroVax™, a Novel Therapeutic TCR Peptide Vaccine for Pediatric Multiple Sclerosis to demonstrate safety & efficacy 12 subjects with pediatric MS

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: 5 Years to 17 Years
* Genders Eligible for Study: Both
* Accepts Healthy Volunteers: No Criteria
* Subject is between 5 and 17 years of age, inclusive
* Clinically diagnosed Pediatric MS
* Definite Pediatric MS by the revised McDonald criteria (2005) (Appendix A), with a pediatric MS course
* Expanded Disability Status Scale (EDSS) <= score 6.5 (Appendix B) Two or more documented clinical relapses of MS in the preceding 24 months OR one documented clinical relapse of MS in the preceding 12 months prior to screening
* Laboratory values within the following limits:

  * Creatinine 1 . 5 x high normal
  * Hemoglobin

Exclusion Criteria:

* Subjects currently prescribed Campath or Lemtrada

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2020-12-31 (Estimated); Primary Completion 2024-11-09 (Estimated); Study Completion 2024-11-09 (Estimated)

PRIMARY OUTCOMES:
The primary clinical endpoints are comparisons of MRI & WBC measurements between the treatment groups | 26 Weeks
  The primary objective is to compare between treatment groups the cumulative number of new gadolinium enhancing (Gd+) lesions on brain MRI & to compare the increases of WBC white blood cell counts in subjects in the treatment groups with Pediatric MS

SECONDARY OUTCOMES:
A Secondary clinical endpoint is the measurement of FOXP3+ expression | 26 Weeks
  Secondary measurements objectives to compare immunologic evaluations increases in FOXP3+ expression between treatment groups
A Secondary clinical endpoint is the measurment of EDSS scores | 26 Weeks
  To compare between treatment groups the Measures of neurologic disability EDSS scores utilizing the Kurtzke scale, Patients will be assessed using the EDSS, a 25-foot timed walk, and a nine-hole peg test assessments at weeks 0, 4, 8, 12, 16, 20 & 26 visit then exit the study.
A Secondary clinical endpoint is the measurement of clinical relapses | 26 Weeks
  To compare the Analysis of clinical relapses between the treatment groups of Pediatric MS subjects at week 26

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Bartholomew, Ph.D, Study Director — Immune Response BioPharma, Inc.
Locations (1):
- CRO, San Diego, California, United States